CLINICAL TRIAL: NCT03219970
Title: An Observational, Non-interventional, Multi-center, Chart Review Study Conducted Among Patients Enrolled in an AZD9291 Early Access Program in Hong Kong, With Locally Advanced/Metastatic EGFR T790M Mutation-positive NSCLC and Prior Exposure to EGFR TKI Therapy.
Brief Title: Efficacy and Safety of Osimertinib for HK Chinese With Metastatic T790M Mutated NSCLC-real World Setting.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00020
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EGFR T790M positive NSCLC patients: Patients with locally advanced/metastatic EGFR T790M positive NSCLC progressed on previous EGFR TKI treatment.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — 80mg oral daily

SUMMARY:
To assess the efficacy of single-agent osimertinib in relation to EGFR T790M mutant allele fraction (AF) in a real-world setting.

DETAILED DESCRIPTION:
This study will assess the efficacy and safety of single-agent osimertinib in patients with locally advanced or metastatic EGFR T790M-positive NSCLC within the context of the early access program in Hong Kong. In particular, osimertinib treatment efficacy will be assessed in the context of the relationship between EGFR T790M mutant AF and survival outcomes, particularly overall survival. In a real-world setting, analysis of overall survival benefit is considered less sensitive to differences in healthcare systems and standards. Other clinical outcomes including response rate (based on physician's judgement) and time to treatment discontinuation (TTD) will be examined. This study will also describe current practice for molecular testing and EGFR mutation profiles in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in AZD9291 Named Patient Program in Hong Kong
* Patients with confirmed advanced (locally advanced (stage IIIB) or metastatic (stage IV)) NSCLC with a positive test result for the EGFR T790M mutation
* Patients who have previously received EGFR TKI therapy or discontinued an EGFR TKI at the time of enrolment in the study
* Provision of written informed consent (for patients alive at the time of study enrolment)
* Documented patients with trackable medical records

Exclusion Criteria:

* Enrolment in studies that prohibit any participation in this non-interventional study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic T790M mutation-positive NSCLC patients progressed or discontinued from previous EGFR TKI treatment.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Association between T790M mutant status and overal survival | Followed up to 2 years after last patient in
  To assess the association of EGFR T790M mutant allele fraction (AF) level with the overall survival (OS) of subjects with advanced/metastatic EGFR T790M-positive NSCLC treated with osimertinib

SECONDARY OUTCOMES:
Overal survival (OS) | Followed up to 2 years after last patient in
  To estimate OS of subjects with advanced/metastatic EGFR T790M-positive NSCLC treated with osimertinib
RR | Follow up within 6 months after last patient in
  To estimate response rate (RR) and disease control rate (DCR) based on physician's judgement, for the overall study population.
TTD | Followed up to 12 months after last patient in
  To estimate time to treatment discontinuation (TTD) of osimertinib for the overall study population, and for subjects with different EGFR mutation status (T790M/Exon 19 del; T790M/L858R)
Adverse event of special interest | Followed up to 12 months after last patient in
  To assess by number of adverse events of special interest which are pre-defined in protocol, as recorded on the case report form.
T790M mutation testing sample | Within 14 days after enrollment date
  To describe what sample or biopsy collected for testing after disease progression on, or discontinuation of, EGFR TKI therapy in the study population
T790M mutation testing platform | Within 14 days after enrollment date
  To describe the characteristics of the methods used for T790M mutation testing after disease progression on, or discontinuation of, EGFR TKI therapy in the study population
EGFR testing mutation subtype | Within 14 days after enrollment date
  To describe the EGFR mutation status of study subjects after disease progression on, or discontinuation of, EGFR TKI therapy
Treatment pattern | Followed up to 2 years after last patient in
  To describe treatment regimens received by study subjects before and after the start of osimertinib therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Siu Hong, Oscar CHAN, Principal Investigator — Pamela Youde Nethersole Eastern Hospital; Kwok Chi LAM, Principal Investigator — Prince of Wales Hospital; Ho Fun, Victor LEE, Principal Investigator — Queen Mary Hospital, Hong Kong; Shi Feng NYAW, Principal Investigator — Tuen Mun Hospital
Locations (4):
- China (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of wales hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160R00020&attachmentIdentifier=1fcc50ba-6690-4e6a-9841-0959d438b831&fileName=D5160R00020_Synopsis.pdf&versionIdentifier=